CLINICAL TRIAL: NCT02438930
Title: Client-Centered Counseling During Routine/Opt-Out HIV-Testing in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan M. Kiene (Other)
Collaborators: Makerere University (Other); National Institute of Mental Health (NIMH) (NIH); Rhode Island Hospital (Other)
Responsible Party: Sponsor-Investigator, Susan M. Kiene, Assistant Professor, UConn Health
Organization: UConn Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SK_UG_K01; K01MH083536 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: HIV; Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing counseling (Experimental): The brief intervention is adapted from the OPTIONS project, which is a brief client-centered risk reduction intervention for HIV-positive patients in clinical care. The OPTIONS intervention content is based upon the IMB model of health behavior change, and uses motivational interviewing techniques to create client-centered discussions in which HIV counselors and patients collaborate to identify patients' HIV transmission risk behaviors and to mutually identify strategies and goals for reducing the patient's risky behavior.
  The brief intervention will be facilitated by health care providers (nurses, lab technicians) specifically trained in the intervention protocol and will consist of 2 brief counseling sessions occurring during the same-day rapid HIV-testing procedure
  Interventions: Behavioral: Motivational interviewing intervention during HIV testing
- Standard of care counseling (Active Comparator): Participants in this study condition will receive standard-of-care counseling that is usually implemented during HIV testing.
  Interventions: Behavioral: Standard-of-care counseling during HIV testing

INTERVENTIONS:
Behavioral: Motivational interviewing intervention during HIV testing
  Arms: Motivational interviewing counseling
Behavioral: Standard-of-care counseling during HIV testing
  Arms: Standard of care counseling

SUMMARY:
This study pilot tests and intervention to help individuals reduce their risk for acquiring or transmitting HIV. The intervention is implemented when people are tested for HIV in an outpatient clinic in rural Uganda. Approximately half of participants will receive the intervention and the other half will receive the usual counseling provided during HIV counseling and testing.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age,
2. have come to the outpatient clinic for a medical concern (e.g., cough, malaria, but not those seeking voluntary HIV-counseling and testing,
3. sexually active within the prior 3-months,
4. not currently pregnant,
5. no confirmed HIV-positive test result prior to the present HIV-test, and
6. live not more than 30km from Gombe Hospital in Uganda (to facilitate follow-up)

Exclusion Criteria:

* less than 18 years of age,
* having come to the clinic seeking voluntary HIV-counseling and testing,
* not sexually active in prior 3 months,
* currently pregnant,
* confirmed prior HIV positive test,
* live more than 30km from the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Sexual risk behavior | 6 months
  Unprotected sex with serodiscordant or unknown HIV status partners

SECONDARY OUTCOMES:
Uptake of partner testing | 6 months
  Partner uptake of HIV testing

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Kiene, PhD, Principal Investigator — UConn Health
Locations (1):
- Gombe Hospital, Gombe, Uganda

REFERENCES:
- [Background] Kiene SM, Sileo K, Wanyenze RK, Lule H, Bateganya MH, Jasperse J, Nantaba H, Jayaratne K. Barriers to and acceptability of provider-initiated HIV testing and counselling and adopting HIV-prevention behaviours in rural Uganda: a qualitative study. J Health Psychol. 2015 Feb;20(2):173-87. doi: 10.1177/1359105313500685. Epub 2013 Sep 20. PMID 24058127